CLINICAL TRIAL: NCT00123006
Title: Cardiovascular and Renal Hemodynamics and the DASH Diet
Brief Title: Effectiveness of the DASH Diet at Reducing High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Paul Conlin, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 229; R01HL077234 (NIH)
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Diseases; Hypertension; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Heart Diseases | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Dietary Approaches to Stop Hypertension (DASH)
  Interventions: Behavioral: Dietary Approaches to Stop Hypertension (DASH)
- 2 (Placebo Comparator): Control diet
  Interventions: Behavioral: Control Diet

INTERVENTIONS:
Behavioral: Dietary Approaches to Stop Hypertension (DASH) — 4 week feeding intervention
  Arms: 1
Behavioral: Control Diet — 4 week feeding intervention
  Arms: 2

SUMMARY:
The purpose of this study is to test the effects of the DASH diet in patients with isolated systolic hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

The study expands upon the findings of the Dietary Approaches to Stop Hypertension (DASH) study, which showed that a dietary pattern emphasizing fruits, vegetables, and low fat dairy products and overall reduced in total and saturated fat significantly lowers blood pressure (BP). The DASH diet is particularly effective in African Americans and in individuals with systolic hypertension. However, it is not known if the DASH diet affects the pathophysiology of the hypertensive process. Preliminary data support the possibility that the DASH diet interrupts the renin-angiotensin system. This raises the intriguing possibility that the DASH diet will favorably impact on cardiovascular and renal hemodynamics in patients with isolated systolic hypertension. Therefore, the central hypothesis of this study is that the DASH diet affects central aortic stiffness, diastolic relaxation, and renal and vascular reactivity to angiotensin II (Ang II) by lowering tissue renin-angiotensin system activity.

DESIGN NARRATIVE:

A randomized, crossover design will be used to compare the DASH diet to a control diet as defined in the original DASH protocol (NEJM 1997; 336:1117). Fifty-five community-dwelling individuals age 20 and older with systolic blood pressure (SBP) 140-179 mmHg and diastolic blood pressure (DBP) less than 90 mmHg will enter a 1-week run-in period eating both the control and DASH diets for 3-4 days each. Following this, participants will begin two 4-week intervention feeding periods receiving either the DASH diet or the control diet in random order. Clinical measurements will be taken at the conclusion of each 4-week feeding period.

Outcome measures: Specific measurements will include peripheral and renal vascular response to Ang II infusions, renal blood flow measured by para-aminohippurate (PAH) clearance, conduit vessel hemodynamics, and tissue Doppler imaging (TDI). At the end of each intervention feeding period, the clinical measurements will be made before and after acute administration of captopril, an angiotensin converting enzyme (ACE) inhibitor.

The study will test whether the DASH diet (1) lowers central aortic stiffness as measured by vascular impedance and carotid-femoral pulse wave velocity; (2) improves diastolic relaxation as measured by early diastolic myocardial velocities across the mitral valve (Ea); (3) vasodilates renal blood flow and enhances vascular responses to Ang II; and (4) affects central aortic stiffness, diastolic relaxation, renal blood flow, and renal and vascular reactivity to Ang II by altering target tissue responsiveness to Ang II similar to ACE inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Isolated systolic hypertension: systolic blood pressure (SBP) in the range of 140-179 mm Hg and diastolic blood pressure (DBP) less than 90 mm Hg
* Body mass index (BMI) less than 40
* Current use of fewer than two blood pressure medications (which will be withdrawn prior to study)

Exclusion Criteria:

* Major concomitant diseases that may include but are not limited to active pulmonary disease within the past 6 months
* History of cardiovascular disorders such as angina, heart attack, heart failure, or stent placement
* Active gastrointestinal disease, including prior gastrointestinal surgery
* Renal disease with serum creatinine greater than 1.5 mg/dl (men) or 1.4 mg/dl (women)
* Insulin-dependent diabetes mellitus
* Current pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-01; Primary Completion 2009-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Changes in central aortic stiffness, diastolic relaxation, renal blood flow,and vascular response to Ang II | Measured at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul R. Conlin, MD, Principal Investigator — Brigham and Women's Hospital

REFERENCES:
- [Derived] Maris SA, Williams JS, Sun B, Brown S, Mitchell GF, Conlin PR. Interactions of the DASH Diet with the Renin-Angiotensin-Aldosterone System. Curr Dev Nutr. 2019 Jul 31;3(9):nzz091. doi: 10.1093/cdn/nzz091. eCollection 2019 Sep. PMID 31528838